CLINICAL TRIAL: NCT03943563
Title: Comparison of Diagnostic Performance of DIXON Sequences With CHESS Sequences by Calculation of the RAMRIS Score in Early Rheumatoid Arthritis
Brief Title: Compare Diagnostic Performance of DIXON &CHESS Sequences Calculating RAMRIS Score in Early Rheumatoid Arthritis.
Acronym: IDEAL PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ideal PR; 2016/24FEV/069 (Other: CEHF)
Record Dates: First submitted 2019-03-19; First posted 2019-05-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Masking Description: None at the time of intervention. At the end of the study, Blind reading without knowledge of the type: Dixon or "classic" sequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single cohort (Other): There is only one cohort where each patient experiment the "classic sequences" as the standard of care and the DIXON sequences for the study.
  Interventions: Diagnostic Test: Dixon sequences acquisition

INTERVENTIONS:
Diagnostic Test: Dixon sequences acquisition — Dixon sequences acquisition

SUMMARY:
In a preliminary MRI study of healthy volunteers's hands investigators showed that the suppression of the fat signal obtained by the Dixon sequences is greater than that obtained by the "classic" CHESS sequences with a better T1-weighted image quality. The investigators goal now is to compare these sequences in the quantification of the inflammatory activity of rheumatoid arthritis by the RAMRIS score. To investigators knowledge, only one study compared those two types of sequence with many limitations including a limited number of patients included.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common chronic inflammatory arthropathy and it mostly affect young women. The MRI sequences currently validated for the joint inflammation assessment are the fat-suppressed sequences produced either by spectral presaturation (CHESS sequences) or by inversion-recovery (STIR = short tau inversion recovery sequence). The presaturation sequences outweigh the STIR sequence due to higher spatial resolution at the expense of sometimes more random saturation of the fat signal. Recently, a third method of suppressing the fat signal (Dixon method) has reappeared thanks to advances in computing power (post-processing). In a preliminary MRI study of the hands of healthy volunteers, the investigators showed that the suppression of the fat signal obtained by the Dixon sequences is greater than that obtained by the "classic" CHESS sequences in T1 and T2 weighting with better quality. image in T1 weighting. This increased performance, particularly in terms of fat suppression, could lead to better detection of PR lesions on MRI.

ELIGIBILITY:
Inclusion Criteria:

* - Rheumatoid arthritis diagnosis for less than 3 years

Exclusion Criteria:

* contraindication to Dotarem contrast injection
* contraindication to MRI due to incompatible implanted material (peacemaker, prosthesis,...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Ramris score | an average of 3 year
  * Calculation of the Rheumatoid Arthritis MRI Scoring System (RAMRIS score) for each sequence by two independent radiologists. RAMRIS is used to evaluate erosions (scale, 0-10, 10 representing the worst situation), edema (scale, 0-3, 3 representing the worst situation), and synovitis (scale, 0-3, 3 representing the worst situation)
  * Blind reading without knowledge of the type of Dixon or "classic" sequence

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium